CLINICAL TRIAL: NCT03439631
Title: ACTION in the OR: Patient Satisfaction With High Efficiency OR Design in Orthopedic Surgery
Brief Title: Patient Satisfaction With Tiered OR Versus Status Quo OR
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's (Other)
Responsible Party: Principal Investigator, Abdelrahman Lawendy, PI, London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 110936
Record Dates: First submitted 2018-02-07; First posted 2018-02-20 (Actual); Last update posted 2023-11-13 (Actual); Status verified 2023-11

CONDITIONS: Surgery

STUDY DESIGN:
Intervention Model Description: Tiered OR set up design will be compared to standard OR set up design as related to patient satisfaction with surgical experience
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Tiered OR Satisfaction (Active Comparator): Patient satisfaction questionnaire with surgical experience in Tiered OR
  Interventions: Other: Patient satisfaction questionnaire
- Status Qou OR satisfaction (Other): Patient satisfaction questionnaire with surgical experience in Tiered OR
  Interventions: Other: Patient satisfaction questionnaire

INTERVENTIONS:
Other: Patient satisfaction questionnaire — Patient satisfaction questionnaire

SUMMARY:
Operating room (OR) costs consume a significant portion of hospital budgets. Standard or "Status Quo" ORs are equipped with the same, fixed set of assigned resources, regardless of case complexity or actual resource requirements. Allocation of resources in standard ORs is the same whether the participant is having heart surgery or bunion removal.

The investigators propose a strategy for OR design and set up wherein resources are carefully matched to procedure complexity as a novel means of healthcare delivery.

This prospective, comparative cohort pilot study will compare two operating room (OR) setup designs. The Tiered OR setup (study intervention) will be an efficiently staffed and equipped OR, geared to the complexity of the surgical procedure. The level of care provided would be equivalent to that of an out-patient day surgery setup. The Status Quo OR setup (control intervention) will be a standard fully equipped, fully staffed OR.

DETAILED DESCRIPTION:
There is an unmet demand for surgical services in Ontario. The situation worsens as the population ages(9). Ontario healthcare costs account for a staggering 40% of the provincial budget(1).Provincial budget deficits mean an influx of healthcare resources are not forthcoming. The aging population costs Ontarians in excess of $2 billion dollars annually(1).

Constrained and overburdened OR resources can result in patients having surgery at night and sometimes surgical procedures being performed by staff not specialized for surgical procedure type(8). Moreover, patient outcomes often decline while they await their surgical date(4, 10-13).

Operating rooms are regarded as an area of intensive resource requirements. With no regard to the complexity of a given procedure or demonstrable resource requirements, ORs are typically managed at critical care levels. This is true for specialized support staff like nurses as well(14). Allocation of resources is not tailored to the individual scenario. This inefficient model of surgical care delivery has been the status quo for decades and the fiscal impact, as well as the challenges this poses to productivity, have taken a toll on hospital budgets and contributed to lengthy provincial wait times for surgical procedures stretching months and even years. For example, according to Health Quality Ontario, the average wait times for elective orthopaedic surgery procedures at London Health Science Center (LHSC) is 96 days to first surgical consultation and an average of 211 days to operating on the patient.

Faced with rising costs in an aging population, the investigators are compelled to find innovative solutions that will allow hospitals to accomplish more with less. These changes are necessary to maintain the standard of Canadian healthcare system and provide timely services in a cost-efficient manner.

Standard or "Status quo" OR set ups are always equipped with the same, fixed set of assigned resources, regardless of case complexity or actual resource requirements. Allocation of resources in standard ORs is the same whether one is having heart surgery or bunion removal.

To challenge these apparent incongruities, the investigators and the hospital pilot tested a tiered strategy for surgical procedures wherein resources were carefully matched to procedure complexity. Preliminary results suggested dramatic improvements in efficiency (up to 35%) and reductions in cost (up to 62%). This Academic Centre Tiered Operating Room strategy (ACTION-in-the-OR) presents a shift from the old, one-size-fits-all OR archetype to a novel, efficient model.

By reducing OR time for minor procedures, the surplus OR time saved could be made available for the more time consuming surgical procedures and for more patients overall. Specialization and standardization has the potential to improve access and quality of care.

This project evaluates an attempt to employ tiered ORs to redistribute finite surgical care resources with orthopedic surgery. While results from a pilot test of high efficiency OR was positive, demonstrating case cost reductions and increased efficiency in OR turnover, longer follow-up, larger sample size, an economic evaluation, and additional high quality evidence is needed to bolster this work.

The investigators propose a prospective, comparative cohort study to evaluate the viability of an altered surgical health care delivery model on participant satisfaction and clinical outcomes as well as economic impact of an innovative healthcare delivery model in orthopedic patients undergoing elective foot and ankle surgery. This project is a portion of a larger proposal which also will examine the impact of tiered OR design on other surgical procedures in arthroplasty and general surgery.

ELIGIBILITY:
Inclusion Criteria:

* • ≥18 years of age

  * No significant co-morbidities preventing outpatient day surgery
  * Undergoing procedures considered a Low Surgical Resource Requirement of relatively short duration with minimal equipment needs (e.g. bunion, revisions, ankle fractures, removal of hardware etc.)
  * Procedures allowing for standardization of equipment and staff

Exclusion Criteria:

* • Refusal to participate

  * Inability to provide informed consent
  * Likely problems maintaining follow-up in the opinion of the investigator
  * Undergoing multiple operative procedures
  * Unable to read/write English even with the aid of an interpreter (for consent and questionnaire completion).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2018-02-28 (Actual); Primary Completion 2023-11-10 (Actual); Study Completion 2023-11-10 (Actual)

PRIMARY OUTCOMES:
Patient surgical Experience Satisfaction survey | 2 weeks post surgery
  patient satisfaction with surgical process
EQ5D- 5L | 2, 6 weeks, 3, 6 months
  change in patient satisfaction with quality of life
NSQIP Patient Reported Surgical Satisfaction Questionnaire | 6 weeks post surgery
  patient satisfaction with surgical process

SECONDARY OUTCOMES:
Resource Utilization Cost Data | baseline to 6 months
  comparison of cost measures between the 2 OR designs

CONTACTS AND LOCATIONS:
Overall Officials: Abdel Lawendy, Principal Investigator — Lawson HRI
Locations (1):
- LHSC, Victoria Hospital, London, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No